CLINICAL TRIAL: NCT06268028
Title: The Effect on the Level of Readiness for Discharge of Discharge Training Given to Primiparous Mothers Having a Cesarean Delivery : A Randomized Controlled Study
Brief Title: Discharge Training Given to Primiparous Mothers Who Had a Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Belma Toptas Acar, Research Assistant Doctor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BELMA TA
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Training
Keywords: Training of discharge; Caesarean section; Primiparous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENT GROUP (Experimental): The individual identification form was first filled out using the face-to-face interview technique. An explanation given regarding filling out the scale and they will be asked to fill it out by self-reporting method under observation. When the mothers in the training group feel good and ready; discharge training gave using the discharge training brochure prepared by the researchers by reviewing the literature. We provided discharge training in the mother's own room and in an average of 30-45 minutes with a one-on-one training method. Mothers asked to fill out the "RHD-NMF" themselves again, close to postnatal discharge.
  Interventions: Behavioral: Training
- CONTROL GROUP (No Intervention): Starting from the first (smallest number) room in the clinic, the individual identification form was filled out initially by face-to-face interview technique for mothers who meet the appropriate conditions and agree to participate in the study, according to the randomization order. An explanation given regarding filling out the scale and they will be asked to fill it out by self-reporting method under observation. Mothers asked to fill out the "RHD-NMF" themselves again, close to postnatal discharge.

INTERVENTIONS:
Behavioral: Training — Discharge training
  Arms: EXPERIMENT GROUP

SUMMARY:
This study aimed to determine the effect of discharge training given to primiparous mothers who gave birth by cesarean section on the level of readiness for discharge.

The research is a pre-test-post-test, randomized controlled experimental study.

DETAILED DESCRIPTION:
The research is a pre-test-post-test, randomized controlled experimental study. To prevent selection bias, participants were included in the training and control groups by applying the randomization method. The sample consisted of a total of 70 women (experimental group: 35 women and control group: 35 women). The study was carried out with women who lying to Obstetrics Clinic of Aydın Gynecology and Children's Diseases Hospital and met the study criteria.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish,
* At least primary school graduate,
* 18 years and over,
* Those who gave birth by cesarean section,
* Primiparous mothers will be included in the research.

Exclusion Criteria:

* Those who have a physical disability (vision, hearing, etc.) that prevents them from taking care of themselves,
* In a risky postpartum period,
* Having a history of chronic disease,
* Those who were hospitalized during pregnancy,
* Those who do not have their baby with them after birth,
* Foreign nationals,
* Mothers with psychiatric diagnoses will not be included in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
A pre-test applied to 70 women who constitute the sample of the research. | 16 weeks
  In the pre-test; The individual introduction form and scale used, and the same scale used for the post-test. Individual Introduction Form: Sociodemographic (Age, educational status, health insurance, etc.) and obstetric characteristics (number of pregnancies, number of miscarriages/abortions etc). (15 questions) (RHD-NMF): Scale that evaluates readiness for hospital discharge according to the mother's perception; It consists of four subscales and a total of 23 items. The lowest score that can be obtained from the scale is '0' and the highest score is '220'.

SECONDARY OUTCOMES:
Apost-test applied to 70 women who constitute the sample of the research. | 16 weeks
  When the mothers in the training group feel good and ready; discharge training was provided using the discharge training brochure prepared by the researchers by reviewing the literature. Discharge training gave one-on-one in the mother's own room, lasting approximately 30-45 minutes. Lectures and question-answer methods used as training techniques. Close to postpartum discharge, mothers in both groups asked to fill out the "RHD-NMF" (post-test) themselves again.

CONTACTS AND LOCATIONS:
Overall Officials: BELMA TOPTAŞ ACAR, Res.assist, Principal Investigator — Res.assist
Locations (1):
- Aydın Maternity and Child Health Hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
OUR STUDY WAS SUPPORTED BY TUBITAK-2209-A UNIVERSITY STUDENTS RESEARCH PROJECTS SUPPORT PROGRAM. OUR DATA COLLECTION PROCESS FİNİSHED.
Supporting Information: CSR
Time Frame: January 10-April 30
Access Criteria: Clinical Study Report (CSR)